CLINICAL TRIAL: NCT07378891
Title: Künstliche Intelligenz (KI)-gestützte Früherkennung Der Diabetischen Retinopathie (FUNDUS-KI)
Brief Title: Artificial-Intelligence-based Early Detection of Diabetic Retinopathy (FUNDUS AI)
Acronym: FUNDUS AI
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 419/2025BO2
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Diabetes (DM); Prediabetes
Keywords: Diabetic retinopathy; Prediabetes; Diabetes; EyeArt
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prediabetes and Diabetes: Participants with prediabetes and diabetes

SUMMARY:
Examination of individuals with prediabetes and established diabetes for early signs of diabetic retinopathy.

DETAILED DESCRIPTION:
Fundus images are acquired and analyzed using an AI algorithm. The fundus images are captured using two devices: a stationary fundus camera (CenterVue DRSplus) and the Optomed Aurora IQ handheld fundus camera. Retinal images are examined using AI-based image analysis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary adults
* Aged between 18 and 80 years
* Understanding of the study explanations and instructions
* Prediabetes (defined by elevated fasting glucose 100-125 mg/dL and/or 2-hour glucose in the oral glucose tolerance test of 140-199 mg/dL and/or HbA1c of 5.7-6.4%)
* manifest diabetes (all types of diabetes according to Ahlqvist)

Exclusion Criteria:

* participants unable to give consent
* Those who do not agree to be informed about incidentally detected pathological findings
* Uncontrolled arterial hypertension (Stage III) despite multiple antihypertensive medications
* Eye diseases that impair the interpretability of the fundus examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients in the University Hospital Tuebingen, volunteers with prediabetes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of retinal changes | Day 1
  Assessment of retinal changes in individuals with prediabetes and diabetes, quantified using an AI algorithm.

SECONDARY OUTCOMES:
Image quality and comparison of the fundus cameras | Day 1
  The automatically assessed image quality and the comparison of stationary and mobile fundus cameras
Influence of clinical parameters on retinal vascular changes | Day 1
  Influence of clinical parameters such as anthropometric measurements (WHR, blood pressure, BMI) and laboratory parameters of glucose and lipid metabolism on retinal vascular changes
Association of medications with the ocular fundus | Day 1
  Association of antidiabetic and lipid-lowering medications with the ocular fundus

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Dep. Diabetology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available